CLINICAL TRIAL: NCT06427746
Title: Accuracy and Implementation of Diagnostic Ability in Stroke in the Pre-Hospital Setting
Brief Title: Enhancing Prehospital Stroke Diagnosis
Acronym: AIPO
Status: Recruiting | Type: Observational
Sponsor: Agenzia Regionale emergenza Urgenza (Other Government)
Responsible Party: Sponsor
Other Study IDs: AREU_A.I.P.O.
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: stroke; video call
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard: stroke diagnosis in the pre-hospital settings, based on the CPSS scale assessed by lay rescuers
  Interventions: Procedure: Standard
- Video call: stroke diagnosis in the pre-hospital settings, based on the CPSS scale assessed by lay rescuers during live video call with the healthcare personnel in EMS dispatch
  Interventions: Procedure: Video call
- Video call + LARIO: stroke diagnosis in the pre-hospital settings, based on the CPSS + LARIO scales assessed by lay rescuers (with specific training on the 2 scales) during live video call with the healthcare personnel in EMS dispatch
  Interventions: Procedure: Video call + LARIO

INTERVENTIONS:
Procedure: Standard — Basic ambulance personnel are trained in the application of the CPSS scale in suspected stroke. The CPSS scale is a tool used to quickly assess stroke severity in pre-hospital settings. It is a three-point scale that takes into account the patient's level of consciousness, facial droop, and arm weakness. If a patient with suspected stroke meets certain criteria, they will be coded as having a suspected stroke by the SOREU. These criteria include having one item in three of the CPSS scale, being of adult age, and being independent at home.
  Groups: Standard
Procedure: Video call — Among the tools already available to improve evaluation of patients rescued in the field, SOREU has video calls between the dispatch room physician and the rescuer in the field. Thus, the rescuer in the field will perform the CPSS during ongoing video call with the dispatch room, allowing the remote evaluation of the patient by the healthcare worker present in the control room, potentially increasing the ability to identify a stroke.
  Groups: Video call
Procedure: Video call + LARIO — LARIO scale's effectiveness in identifying patients with ischemic stroke caused by a large vessel occlusion in the anterior cerebral circulation. The anterior cerebral circulation supplies blood to the front and upper parts of the brain. Occlusion of a large vessel in this area can lead to a severe stroke. Rescuer in the field will perform the CPSS and the LARIO during ongoing video call with the dispatch room, allowing the remote evaluation of the patient by the healthcare worker present in the control room.
  Groups: Video call + LARIO

SUMMARY:
Current American Heart Association Guidelines recommend that stroke patients be promptly rescued and identified so that the accepting hospital can be alerted and prepared to receive and treat them promptly. It is also recommend that stroke identification be performed using validated and standardized assessment scales. This study aims to analyze the possibility to increase the correct identification of stroke patients after implementation of several new operative procedures by the emergency medical service (EMS) of the metropolitan area of Milan (SOREU). The interventions adopted include:

1. the evaluation of patients with suspected stroke via video call between the lay rescue personnel and the dispatch healthcare personnel
2. the training of lay rescue personnel, operating in the metropolitan area, aimed at implementing the application of the Cincinnati Prehospital Stroke Scale (CPSS) scale and to expand the neurological examination with the addiction of the Large ARtery Intracranial Occlusion Stroke Scale (LARIO) in the clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* suspected stroke
* rescued by basic life support vehicle
* consciousness
* informed consent

Exclusion Criteria:

* age < 18 years
* rescued by an advanced life support vehicle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in the prehospital setting with suspected ischemic stroke rescued by the emergency medical service in the Milan metropolitan area
Sampling Method: Probability Sample
Enrollment: 2197 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of prehospital stroke diagnosis | within 2 hours from hospital admission
  Evaluate if the use of the video call with or without the assessment of the LARIO scale, between the prehospital lay rescuer and the medical dispatch improve the identification of stroke patients in comparison to the only CPSS scale evaluated by the lay rescuer. The diagnosis accuracy is evaluated by confirmation of stroke at the cerebral angio-CT scan

SECONDARY OUTCOMES:
Accuracy of the Large ARtery Intracranial Occlusion (LARIO) scale to identify a stroke with occlusion of a large vessels | within 2 hours from hospital admission
  LARIO is a stroke scale is a simple 5-item clinical scale that can be used to predict the presence of large vessel occlusion (LVO) in patients with acute ischemic stroke. A large vessel of the anterior cerebral circulation is defined as occlusion of the intracranial segment of the internal carotid artery, anterior cerebral artery segments A1 and A2, and middle cerebral artery segments M1 and M2. Final diagnosis is based on the cerebral angio CT scan
incidence of hemorrhagic stroke | within 2 hours hospital admission
  incidence of hemorrhagic stroke among patients identified as stroke patients. Diagnosis is based on the results of the cerebral CT

CONTACTS AND LOCATIONS:
Overall Officials: Anna Coppo, MD, Principal Investigator — AREU
Locations (1):
- SOREU Metropolitana, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided